CLINICAL TRIAL: NCT06409143
Title: Neural Mechanisms and Augmented Efficacy of High-definition Transcranial Electrical Stimulation on Upper-extremity Function in Patients With Subacute Stroke
Brief Title: High-definition Transcranial Electrical Stimulation for Upper Extremity Rehabilitation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 202309053DINB
Record Dates: First submitted 2024-05-07; First posted 2024-05-10 (Actual); Last update posted 2024-08-16 (Actual); Status verified 2024-05

CONDITIONS: Stroke
Keywords: Stroke; High-Definition Transcranial Electrical Stimulation; Upper-limb rehabilitation; Transcranial electrical stimulation; Neuroplasticity
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Excitatory stimulation on the affected hemisphere & UE rehabilitation (Experimental): 10 minutes sham inhibitory HD-tES over the unaffected hemisphere's M1 followed by 10 minutes of excitatory HD-tES over the affected hemisphere's M1, combined with upper extremity rehabilitation of affected side.
  Interventions: Device: HD-tES; Other: UE rehabilitation
- Inhibitory stimulation on the unaffected hemisphere & UE rehabilitation (Experimental): 10-minute active inhibitory HD-tES over the unaffected hemisphere's M1 followed by 10 minutes of sham excitatory HD-tES over the affected hemisphere's M1, combined with upper extremity rehabilitation of affected side.
  Interventions: Device: HD-tES; Other: UE rehabilitation
- Simultaneous bilateral stimulation & UE rehabilitation (Experimental): Combined with upper extremity rehabilitation of affected side.
  Interventions: Device: HD-tES; Device: HD-tES (Bilateral)
- Sham stimulation& UE rehabilitation (Sham Comparator): The sham control group will receive sham HD-tCES combined with upper extremity rehabilitation of affected side.
  Interventions: Device: Sham HD-tES; Other: UE rehabilitation

INTERVENTIONS:
Device: HD-tES — The intensity of HD-tES is set at 2 mA, the current intensity ramps up to 2 mA within 5 seconds, remains at 2 mA for 10 minutes, and then ramps down to zero within 5 seconds. For the sham stimulation, the current intensity ramps up and down at the first and last 10 seconds, with the remaining 10 minutes set at 0 mA. The inhibitory and excitatory waveform will be selected based on results of sub-project 1.
  Arms: Excitatory stimulation on the affected hemisphere & UE rehabilitation; Inhibitory stimulation on the unaffected hemisphere & UE rehabilitation; Simultaneous bilateral stimulation & UE rehabilitation
Device: Sham HD-tES — The intensity of HD-tES is set at 2 mA, the current intensity ramps up to 2 mA within 5 seconds, remains at 2 mA for 10 minutes, and then ramps down to zero within 5 seconds. For the sham stimulation, the current intensity ramps up and down at the first and last 10 seconds, with the remaining 10 minutes set at 0 mA. The inhibitory and excitatory waveform will be selected based on results of sub-project 1.
  Arms: Sham stimulation& UE rehabilitation
Other: UE rehabilitation — Upper extremity rehabilitation programs will be selected and graded in accordance with each patient's upper extremity function and specific aims of activities of daily living. Upper extremity rehabilitation will be provided for 60 minutes each time, 5 times a week, lasting for 3 weeks.
  Arms: Excitatory stimulation on the affected hemisphere & UE rehabilitation; Inhibitory stimulation on the unaffected hemisphere & UE rehabilitation; Sham stimulation& UE rehabilitation
Device: HD-tES (Bilateral) — The intensity of HD-tES is set at 2 mA, the current intensity ramps up to 2 mA within 5 seconds, remains at 2 mA for 10 minutes, and then ramps down to zero within 5 seconds.
  Arms: Simultaneous bilateral stimulation & UE rehabilitation

SUMMARY:
Upper limb hemiparesis is the most common sequelae in patients, severely impacting their independence and quality of life. Transcranial electrical stimulation (tCES) is a non-invasive and safe treatment, which uses a low direct current or alternating current to change the excitability of the cerebral cortex. It can induces long-term potentiation-like or long-term depression-like effects, thereby modulating the cortical excitability. In recent years, researchers have developed high-definition (HD) devices, which integrate high definition ring electrode configurations and incorporate direct current with theta burst stimulation waveforms. Diverging from traditional transcranial direct current stimulation (tDCS), which applies weak currents (0.5-2 mA) through two large sponge electrodes (25~35 cm^2) externally to the scalp for widespread non-specific cortical stimulation, HD-tES employs an array of small-area electrodes (1 cm^2) to control current distribution over localized cortical regions, thereby enhancing spatial accuracy. However, there is a lack of studies validating the optimal waveform for HD-tES, as well as clinical evidence in subacute stroke populations. The optimal unilateral versus bilateral stimulation modes and their neurological mechanisms for stroke rehabilitation also remain uncertain.

DETAILED DESCRIPTION:
This project comprises two sub-projects:

1. Investigation of Neuromodulatory Effects of Stimulation Waveforms and Optimal Stimulation Waveform for Patients with Stroke : a crossover trial will compare the effects of seven high-definition transcranial electrical stimulation (HD-tES) waveforms on neural excitatory or inhibitory activity in healthy adults. These waveforms include three excitatory wave forms (anodal direct current (aDC), intermittent theta burst stimulation (iTBS), and a combination of aDC and iTBS (aDC+iTBS)) and three inhibitory wave forms (cathodal direct current (cDC), continuous theta burst stimulation (cTBS), and a combination of cDC and cTBS (cDC+cTBS)), along with a sham stimulation condition. Changes in cortical excitability over a 2-hour period before and after stimulation will be tracked.

   Validation of the optimal stimulation waveform for patients with stroke will be conducted through a crossover trial comparing three excitatory HD-tES waveforms for enhancing affected brain activity and three inhibitory HD-tES waveforms for reducing activity in the unaffected hemisphere. Changes in cortical excitability over a 2-hour period before and after stimulation will be monitored.
2. Exploration of the Effects of Unilateral and Bilateral HD-tES in Patients with Subacute Stroke: A triple-blind randomized controlled trial will be conducted to compare four neuromodulatory modes combined with conventional upper limb rehabilitation on brain activity and upper limb function in patients with subacute stroke. These modes include excitatory stimulation on the affected hemisphere (based on results from sub-project one, choosing from aDC, iTBS, or aDC+iTBS), inhibitory stimulation on the unaffected hemisphere (based on results from sub-project one, choosing from cDC, cTBS, or cDC+cTBS), simultaneous bilateral stimulation, and sham stimulation.

The primary outcome will focus on upper limb functional activity and upper limb motor function, with other indicators serving as secondary outcomes.

ELIGIBILITY:
Inclusion Criteria:

- Sub-Project 1 (Healthy)

1. Adults aged 18 and above.
2. Confirmed right-handedness using the Edinburgh Handedness Inventory.

Sub-Project 1 (Post-stroke patients)

1. Aged 18 and above.
2. Diagnosed with stroke.
3. Post-stroke for more than 6 months.
4. Unilateral hemiparesis.

Sub-Project 2 (Subacute-stroke patients)

1. Aged 18 and above.
2. Diagnosed with stroke.
3. Stroke occurred between 7 days to 6 months ago.
4. Unilateral hemiparesis.
5. Degree of recovery for proximal and distal movements of the affected upper limb is Brunnstrom stage III to V.
6. No severe muscle spasticity in any segments of the affected upper limb (Modified Ashworth Scale ≤ 2).

Exclusion Criteria:

- Sub-Project 1 (Healthy)

1. History of neurological disorders (e.g., stroke, brain tumor, epilepsy), psychiatric disorders (e.g., substance abuse, major depression, schizophrenia, bipolar disorder), or musculoskeletal disorders of the upper limb.
2. Contraindications to transcranial electrical stimulation, including history of epilepsy, atrial fibrillation, presence of metal implants, cardiac pacemakers, convexity skull defects, or increased intracranial pressure.
3. Skin allergies, contact dermatitis, abnormal pain, hypersensitivity to pain, wounds, or ulcers on the head.
4. Participation in other invasive or non-invasive brain stimulation research studies.
5. Pregnancy or lactating women. (If female, must be postmenopausal or surgically sterilized. Fertile women must have a negative pregnancy test result. Fertile female patients engaging in heterosexual intercourse, as well as fertile male patients with fertile female partners, must agree to use effective contraception during the trial period and for 4 months after the last dose of the investigational drug, such as oral contraceptives, dual barrier methods, intrauterine devices, or abstain from sexual intercourse during this period; non-fertile women are those who have undergone bilateral oophorectomy or are postmenopausal.)
6. History of alcohol or substance abuse.
7. Damaged skin at the stimulation site, electrode contact, or device wearing site.
8. Long-term use of central nervous system affecting medications (such as antidepressants, sedatives) or other medications that may affect seizure threshold.
9. Other conditions deemed unsuitable for transcranial electrical or magnetic stimulation by a physician.
10. Affiliation with any research institution/execution unit (e.g., students from NTU, Taipei Medical University).

Sub-Project 1 (Post-stroke patients)

1. Contraindications to transcranial electrical stimulation include a history of epilepsy, atrial fibrillation, presence of metal implants, cardiac pacemakers, convexity skull defects, or increased intracranial pressure.
2. Skin allergies, contact dermatitis, abnormal pain, hypersensitivity to pain, wounds, or ulcers on the head.
3. Severe neurological or psychiatric disorders other than stroke (such as major depression, schizophrenia, substance abuse, organic brain diseases, Parkinson's disease, brain tumors).
4. Use of medications that may lower the seizure threshold.
5. Undergoing other invasive or non-invasive brain stimulation therapies.
6. Pregnancy or lactating women. (If female, must be postmenopausal or surgically sterilized. Fertile women must have a negative pregnancy test result. Fertile female patients engaging in heterosexual intercourse, as well as fertile male patients with fertile female partners, must agree to use effective contraception during the trial period and for 4 months after the last dose of the investigational drug, such as oral contraceptives, dual barrier methods, intrauterine devices, or abstain from sexual intercourse during this period; non-fertile women are those who have undergone bilateral oophorectomy or are postmenopausal.)
7. History of alcohol or substance abuse.
8. Damaged skin at the stimulation site, electrode contact, or device wearing site.
9. Long-term use of central nervous system affecting medications (such as antidepressants, sedatives) or other medications that may affect seizure threshold.
10. Other conditions deemed unsuitable for transcranial electrical or magnetic stimulation by a physician.

Sub-Project 2 (Subacute-stroke patients)

1. Contraindications to transcranial electrical stimulation include a history of epilepsy, atrial fibrillation, presence of metal implants, cardiac pacemakers, convexity skull defects, or increased intracranial pressure.
2. Skin allergies, contact dermatitis, abnormal pain, hypersensitivity to pain, wounds, or ulcers on the head.
3. Severe neurological or psychiatric disorders other than stroke (such as major depression, schizophrenia, substance abuse, organic brain diseases, Parkinson's disease, brain tumors).
4. Use of medications that may lower the seizure threshold.
5. Other muscle and joint problems affecting upper limb function, such as joint contractures, rheumatoid arthritis, myositis ossificans.
6. Severe cognitive impairment or receptive or global aphasia making it difficult to understand instructions.
7. Hemineglect (including visual, auditory, or sensory neglect).
8. Undergoing other invasive or non-invasive brain stimulation therapies.
9. Pregnancy or lactating women. (If female, must be postmenopausal or surgically sterilized. Fertile women must have a negative pregnancy test result. Fertile female patients engaging in heterosexual intercourse, as well as fertile male patients with fertile female partners, must agree to use effective contraception during the trial period and for 4 months after the last dose of the investigational drug, such as oral contraceptives, dual barrier methods, intrauterine devices, or abstain from sexual intercourse during this period; non-fertile women are those who have undergone bilateral oophorectomy or are postmenopausal.)
10. History of alcohol or substance abuse.
11. Damaged skin at the stimulation site, electrode contact, or device wearing site.
12. Long-term use of central nervous system affecting medications (such as antidepressants, sedatives) or other medications that may affect seizure threshold.
13. Other conditions deemed unsuitable for transcranial electrical or magnetic stimulation by a physician.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 152 (Estimated)
Dates: Start 2024-08-15 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
Pre- and 3-month change in motor function of the upper limbs assessed by Fugl-Meyer Assessment of Upper Extremity (FMA-UE) | Baseline (within 7 days ahead to the 1st intervention session), after 3-week intervention (within 7 days after the last intervention session), follow up (3-month after post-test)
  The FMA-UE assesses motor functioning of upper extremity. Each movement is estimated by a 3-point scale (0-1-2). The total score of the FMA-UE is 66, and a higher score indicates that the patient has better movement ability.
Pre- and 3-month change in motor function of the upper limbs assessed by Action Research Arm Test (ARAT) | Baseline (within 7 days ahead to the 1st intervention session), after 3-week intervention (within 7 days after the last intervention session), follow up (3-month after post-test)
  ARAT consists of 19 items,including grasp (6 items), grip (6 items), pinch (6 items), and gross movement (3 items). Each item is scored on a scale of 0-1-2-3, where 0 indicates the complete inability to perform the movement, 1 indicates partial completion of the movement, 2 indicates independent completion of the movement but with excessive time or difficulty, and 3 indicates a movement pattern that is roughly normal. The total score ranges from 0 to 57, with higher scores indicating better upper limb functional ability.

SECONDARY OUTCOMES:
Pre- and 3-month change in motor function of the upper limbs assessed by Modified Ashworth Scale (MAS) | Baseline (within 7 days ahead to the 1st intervention session), after 3-week intervention (within 7 days after the last intervention session), follow up (3-month after post-test)
  The MAS is commonly used in clinical practice for grading spasticity. The MAS is rated on a 6-point scale (0, 1, 1+, 2, 3, 4), and a higher score indicates that the patient has higher muscle tension. The muscles being assessed include shoulder abductor, elbow flexor, elbow extensor, wrist flexor, and finger flexor.
Pre- and 3-month change in sensory function of the upper limbs assessed by Rivermead Assessment of Somatosensory Performance (RASP) | Baseline (within 7 days ahead to the 1st intervention session), after 3-week intervention (within 7 days after the last intervention session), follow up (3-month after post-test)
  There are a total of 33 items, among which 5 items assess facial and upper and lower limb tactile discrimination, 5 items assess facial and upper and lower limb pressure sensation, 5 items assess facial and upper and lower limb tactile localization, 2 items assess facial and hand sensory extinction, 1 item assesses finger two-point discrimination, 5 items assess facial and upper and lower limb temperature sensation, 5 items assess upper and lower limb proprioception, and 5 items assess upper and lower limb kinesthesia. Each item is tested 6-9 times, and scores are calculated based on the number of correct responses, with higher scores indicating better somatosensory function.
Pre- and 3-month change in used and quality of affected extremity assessed by Motor Activity Log (MAL) | Baseline (within 7 days ahead to the 1st intervention session), after 3-week intervention (within 7 days after the last intervention session), follow up (3-month after post-test)
  The questionnaire assesses the frequency and quality of use of the affected upper limb in daily activities for stroke or brain injury patients with hemiparesis. There are a total of 30 items representing common daily activities, with each item scored on a scale of 0-5. A score of 0 indicates no use of the affected side, while a score of 5 indicates the same frequency and quality of use as before the onset of the condition. The total score is calculated as the average score across the 30 items, with higher scores indicating better frequency of use or quality of movement of the affected upper limb.
Pre- and 3-month change in quality of life assessed by Stroke Impact Scale 3.0 (ML-SIS) | Baseline (within 7 days ahead to the 1st intervention session), after 3-week intervention (within 7 days after the last intervention session), follow up (3-month after post-test)
  The ML-SIS questionnaire comprises 28 items designed to evaluate different aspects of stroke patients' quality of life. These aspects include muscle strength, memory, emotional status, communication ability, activities of daily living (ADL), mobility, hand function, and social participation. Each item within these categories is scored on a scale from 1 to 5, with higher scores indicating a better quality of life.This comprehensive assessment tool provides insights into various domains of stroke survivors' well-being.
Everytime report for the incidence of treatment-emergent adverse events [safety and tolerability] | Within 10 minutes after each intervention session (a total of 15 sessions, 5 sessions/week, lasting 3 weeks)
  Immediately after each HD-tES stimulation, the patient will be questioned about eventual side effect

OTHER OUTCOMES:
Pre- and 3-month change in cerebral hemodynamic assessed by functional near-infrared spectroscopy (fNIRS) | During each intervention session (a total of 15 sessions, 5 sessions/week, lasting 3 weeks)
  The researchers will utilize the NIRSport 2 functional near-infrared spectroscopy (fNIRS) system to collect cerebral hemodynamic parameters in the sensorimotor cortex regions bilaterally of the subjects. Aimed to estimate changes in functional activation and connectivity of corresponding brain areas before and after intervention. The fNIRS system employs two wavelengths, 760 nm and 850 nm, of near-infrared light.
  fNIRS involves an initial 5-minute resting state measurement, during which the subjects are instructed to sit with eyes open, remain as still as possible, maintain a calm and relaxed emotional state, and try not to think about anything. Subsequently, task-induced brain activation fNIRS measurements will be initiated, wherein subjects will perform a fist-clenching task for 20 seconds followed by a 30-second rest period before proceeding to the next round of the task. This cycle will be repeated for a total of 8 rounds.
Pre- and 3-month change in neuronal activation assessed by motor evoked potential, MEP | Baseline (within 7 days ahead to the 1st intervention session), after 3-week intervention (within 7 days after the last intervention session), follow up (3-month after post-test)
  MEP (Motor Evoked Potential) is elicited by single-pulse transcranial magnetic stimulation (TMS) targeting the first dorsal interossei (FDI) muscle, corresponding to the specific area of the brain's motor cortex. During the first week, subjects will undergo M1 hand motor hotspot localization before receiving HD-tES.
  Each week before HD-tES, rMT will be measured by delivering ten magnetic stimuli, with at least five eliciting MEPs of 50 µV or more in the FDI muscle. The stimulation intensity at this point is recorded as rMT, representing the minimum intensity required to evoke a motor response in the resting muscle, with smaller values indicating higher neural activity.Participants will undergo MEP measurements bilaterally at 0, 10, 20, 30, 40, 50, 60, 90, and 120 minutes before and after HD-tES. Additionally, at the end of the session, MEPs will be measured using a stimulation intensity of 120% of rMT, repeated ten times, with the average amplitude representing MEP.

CONTACTS AND LOCATIONS:
Locations (3):
- Taiwan (3):
  - New Taipei City Tucheng Hospital, New Taipei City
  - National Taiwan University Hospital, Taipei
  - Taipei Medical University Hospital, Taipei